CLINICAL TRIAL: NCT00067717
Title: Placebo Effects in Distance Healing of Wounds
Brief Title: Distance Healing in Wound Healing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Marilyn Schlitz, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21AT001437 (NIH); R21AT001437 (NIH); SchlitzMJ
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Breast Reconstruction Surgery
Keywords: breast reconstruction surgery; prayer; distance healing; wound healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Distant Healing (Experimental): This group received distant healing but was blinded to the condition.
  Interventions: Behavioral: Distance healing
- Non-blinded Distant Healing (Placebo Comparator): This group received the distant healing intervention and was called every day they were receiving to be told they were receiving it, therefore enhancing expectancy.
  Interventions: Behavioral: Distance healing
- Blinded Control (No Intervention): This group was blinded to the intervention condition and did not receive any distant healing.

INTERVENTIONS:
Behavioral: Distance healing
  Arms: Distant Healing; Non-blinded Distant Healing

SUMMARY:
This trial examines the impact of patients' knowledge of an experienced distant healer's efforts to heal them on measures of wound healing, psychosocial functioning, and physiological symptoms after plastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing major plastic surgery (> 2 hours in length)
* Health status is excellent with no systemic disease, no limitation on activity, no danger of death or disease of one body system, well-controlled underlying disease

Exclusion Criteria:

* Remove history of breast or other cancers
* History of radiation therapy to the abdomen or any radiation within the past three months
* Non-English speaking
* Unable or unwilling to fill out questionnaires
* Current smoker
* Morbid obesity
* Circulatory inadequacies (i.e., diabetes, hypovolemia)
* Nutritional deficits as evidenced by neutropenia (WBC <2500/ml) or hypoalbuminemia (albumin <3.3mmg/dl) / chart review

Ages: 34 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2003-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Collagen deposition in a surrogate wound | 8 days

SECONDARY OUTCOMES:
POMS normalized mood scores | 8 days
  Compared from baseline to end of distant healing period

OTHER OUTCOMES:
SF-36 Mental Composite Score | 8 days
SF-36 Physical Composite Score | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn J Schlitz, PhD, Principal Investigator — California Pacific Medical Center
Locations (1):
- Complementary Medicine Research Institute, San Francisco, California, United States

REFERENCES:
- [Background] Schlitz M, Hopf HW, Eskenazi L, Vieten C, Radin D. Distant healing of surgical wounds: an exploratory study. Explore (NY). 2012 Jul-Aug;8(4):223-30. doi: 10.1016/j.explore.2012.04.004. PMID 22742672